CLINICAL TRIAL: NCT02972125
Title: A Single-Center, Open-Label, Randomized, Single-Oral Dose, 2-Way Cross-Over Study to Investigate the Bioequivalence Between Lacosamide Tablet and Dry Syrup in Healthy Male Japanese Subjects
Brief Title: A Study to Demonstrate the Bioequivalence of Lacosamide Tablets and Dry Syrup in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EP0059; 2016-002462-31 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Lacosamide; Bioequivalence; Dry Syrup
MeSH Terms: interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A - B (Experimental): Single administration of the reference drug (Treatment A, a single dose of Lacosamide (LCM) 100 mg tablet), followed by a Wash-Out Period of at least 7 days and a single administration of the test drug (Treatment B, a single dose of LCM 100 mg given as dry syrup).
  Interventions: Drug: Lacosamide (LCM) tablet; Drug: Lacosamide (LCM) dry syrup
- Treatment B - A (Experimental): Single administration of the test drug (Treatment B, a single dose of LCM 100 mg given as dry syrup), followed by a Wash-Out Period of at least 7 days and a single administration of the reference drug (Treatment A, a single dose of Lacosamide (LCM) 100 mg tablet).
  Interventions: Drug: Lacosamide (LCM) tablet; Drug: Lacosamide (LCM) dry syrup

INTERVENTIONS:
Drug: Lacosamide (LCM) tablet — Treatment A: Single dose of Lacosamide (LCM) 100 mg tablet
Drug: Lacosamide (LCM) dry syrup — Treatment B: Single dose of Lacosamide (LCM) 100 mg given as dry syrup

SUMMARY:
This is a study designed to demonstrate the Bioequivalence between Lacosamide (LCM) Tablet and Dry Syrup in Healthy Male Japanese Subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject is male and between 20 and 55 years of age (inclusive)
* Subject is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (a subject has all 4 Japanese grandparents born in Japan)
* Male subject confirms that when having sexual intercourse with a woman of childbearing potential, he will use condoms during the study and 1 week after the last dose of study drug

Exclusion Criteria:

* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study.
* Subject has clinically relevant out-of-range values for hematology, and serum chemistry, or urinalysis variables at the Screening Visit.
* Subject has any clinically significant abnormal physical examination (Screening Visit or Day -1) and vital signs (Screening Visit).
* Subject has any clinically relevant ECG finding at the Screening Visit.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
Area under the curve from 0 to time of last quantifiable concentration (AUC(0-t)) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing

SECONDARY OUTCOMES:
Area under the curve from zero up to infinity (AUC) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
Apparent total body clearance (CL/F) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
Apparent volume of distribution (Vz/F) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
Mean residence time (MRT) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
Time of observed Cmax (tmax) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
Terminal elimination half-life (t1/2) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing
First order terminal elimination rate constant (Lambda z) | Blood samples are collected at predose and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Ep0059 001, London, United Kingdom